CLINICAL TRIAL: NCT03387020
Title: A Phase I and Surgical Study of Ribociclib and Everolimus (RAD001) in Children With Recurrent or Refractory Malignant Brain Tumors
Brief Title: Ribociclib and Everolimus in Treating Children With Recurrent or Refractory Malignant Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBTC-050; NCI-2017-02079 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PBTC-050 (Other: Pediatric Brain Tumor Consortium); PBTC-050 (Other: CTEP); UM1CA081457 (NIH)
Record Dates: First submitted 2017-12-05; First posted 2017-12-29 (Actual); Results first posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: CNS Embryonal Tumor, Not Otherwise Specified; Malignant Glioma; Recurrent Atypical Teratoid/Rhabdoid Tumor; Recurrent Childhood Ependymoma; Recurrent Diffuse Intrinsic Pontine Glioma; Recurrent Medulloblastoma; Refractory Diffuse Intrinsic Pontine Glioma
MeSH Terms: conditions — Glioma; Rhabdoid Tumor; Familial ependymoma; Diffuse Intrinsic Pontine Glioma; Medulloblastoma | interventions — Everolimus; ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ribociclib, everolimus) (Experimental): Patients receive ribociclib PO QD on days 1-21 of course 1 and subsequent courses and days 2-21 of course 2, and everolimus PO QD on days 3-28 of course 1 and days 1-28 of subsequent courses. Patients who are undergoing surgery also receive ribociclib PO QD on days 7-10 before surgery. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity. Patients with stable disease after 13 courses may continue receiving ribociclib and everolimus every 28 days for up to 13 additional courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Everolimus; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Ribociclib

INTERVENTIONS:
Drug: Everolimus — Given PO
  Other Names: 42-O-(2-Hydroxy)ethyl Rapamycin; Afinitor; Certican; RAD 001; RAD001; Votubia; Zortress
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Ribociclib — Given PO
  Other Names: Kisqali; LEE-011; LEE011

SUMMARY:
This phase I trial studies the side effects and best dose of ribociclib and everolimus and to see how well they work in treating patients with malignant brain tumors that have come back or do not respond to treatment. Ribociclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as everolimus, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ribociclib and everolimus may work better at treating malignant brain tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and/or the recommended phase II dose (RP2D) of ribociclib and everolimus in children with refractory or recurrent central nervous system (CNS) tumors. (Phase I) II. To describe the toxicity profile and define the dose-limiting toxicities (DLTs) of ribociclib and everolimus in children with refractory or recurrent CNS tumors. (Phase I) III. To characterize the pharmacokinetics of ribociclib and everolimus in children with refractory or recurrent CNS tumors, and the potential for drug-drug interactions between the two compounds in this population. (Phase I) IV. To characterize ribociclib concentrations in tumor, and plasma in children with refractory or recurrent CNS malignancies undergoing neurosurgical procedures. (Surgical Study)

SECONDARY OBJECTIVES:

I. To describe the response rate of relapsed and refractory malignant brain tumors to ribociclib and everolimus in the context of a phase I study. (Phase I) II. To explore the effect of ribociclib treatment on Ki-67 by immunohistochemistry (IHC) by comparing archival and post-treatment tumor tissue. (Surgical Study)

TERTIARY OBJECTIVES:

I. To increase knowledge of the genomic landscape of treatment-refractory pediatric CNS tumors, including mechanisms of resistance and response.

OUTLINE: This is a dose-escalation study.

Patients receive ribociclib orally (PO) once daily (QD) on days 1-21 of course 1 and subsequent courses and days 2-21 of course 2, and everolimus PO QD on days 3-28 of course 1 and days 1-28 of subsequent courses. Patients who are undergoing surgery also receive ribociclib PO QD on days 7-10 before surgery. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity. Patients with stable disease after 13 courses may continue receiving ribociclib and everolimus every 28 days for up to 13 additional courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* ELIGIBILITY FOR SCREENING
* Patients with a histologically confirmed diagnosis of high-grade glioma (HGG), medulloblastoma, CNS embryonal tumor (not otherwise specified [NOS]), ependymoma, or atypical teratoid rhabdoid tumor (ATRT) that is recurrent, progressive or refractory
* Patients with recurrent diffuse intrinsic pontine glioma (DIPG) with typical radiographic appearance who have undergone biopsy are eligible provided there is histologic confirmation of malignant glioma World Health Organization (WHO) II-IV; Rb1 screening for these patients is required only if adequate tissue is available
* Patients with recurrent brainstem tumors with an atypical presentation who have undergone biopsy are eligible provided there is histologic confirmation of malignant glioma WHO II-IV; these patients must undergo Rb1 screening; these patients must have radiographic evidence of progression
* Patients with secondary malignant gliomas will be eligible for this study but should conform to all other eligibility requirements; patients with low-grade gliomas are excluded
* Formalin fixed paraffin embedded tumor tissue (preferably from the most recent recurrence) must be available to assess Rb1 protein status prior to enrollment on phase I or surgical study; if the subject has results from prior Rb1 IHC testing in a Clinical Laboratory Improvement Act (CLIA)-certified laboratory the requirement for screening to assess Rb1 protein status is waived
* Patients with recurrent diffuse intrinsic brain stem glioma (DIPG) that has an atypical presentation must also submit the tumor tissue for Rb1 protein status confirmation or provide previous testing results from a CLIA certified laboratory; patients who have been biopsied for atypical DIPG but do not have sufficient tissue for Rb1 screening are not eligible
* Body surface area (BSA)

  * Patients enrolled on dose level -1 must have BSA >= 0.55m^2
  * Patients enrolled on dose level -0.5 must have BSA >= 0.75m^2
  * Patients enrolled on dose level 0 must have BSA >= 0.55m^2
  * Patients enrolled on dose level 1 must have BSA >= 0.75m^2
  * Patients enrolled on dose level 2 and 3 must have BSA >= 0.45m^2
* Patients who are candidates for enrollment for the phase I or surgical studies must sign a screening consent and provide pre-trial tumor material for Rb1 testing unless testing is not needed due to diagnosis or the availability of prior Rb1 IHC results; the screening consent is to be obtained according to institutional guidelines
* Patients screened for this trial should be expected to meet the criteria for treatment
* PRIOR TO STUDY ENROLLMENT
* PHASE I (STRATUM 1): Patient has intact Rb1 protein confirmed either from previous results or screened tissue; all testing must be performed in a CLIA certified laboratory; DIPG patients with radiographically typical appearance will be waived from this requirement
* PHASE I (STRATUM 1): Patients with a histologically confirmed diagnosis of a primary CNS tumor that is recurrent, progressive, or refractory; all tumors must have histologic verification of HGG, medulloblastoma, CNS embryonal tumor (NOS), ependymoma, or ATRT; patients with low-grade gliomas are excluded
* PHASE I (STRATUM 1): Patients with progressive DIPG, as defined by progressive neurologic abnormalities or worsening neurologic status not explained by causes unrelated to tumor progression (e.g., anticonvulsant or corticosteroid toxicity wean, electrolyte disturbances, sepsis, hyperglycemia, etc.), OR an increase in the bi-dimensional measurement, taking as a reference the smallest disease measurement recorded since last treatment, OR the appearance of a new tumor lesion since diagnosis

  * Please note:

    * Patients with a radiographically typical DIPG, defined as a tumor with a pontine epicenter and diffuse involvement of more than 2/3 of the pons, are eligible without histologic confirmation
    * Patients with pontine lesions that do not meet these radiographic criteria will be eligible if there is histologic confirmation of malignant glioma WHO II-IV. These patients must have radiographic evidence of progression
* SURGICAL STUDY (STRATUM 2): Patients must have recurrent or refractory disease with a histological diagnosis at either the time of diagnosis or at the time of recurrence of one of the following:

  * HGG
  * Medulloblastoma,
  * CNS embryonal tumor (NOS),
  * Ependymoma, or
  * ATRT
* SURGICAL STUDY (STRATUM 2): Patients for whom surgical intervention is clinically indicated (gross total resection or sub-total resection) at recurrence and are amenable to receiving ribociclib for 7 ? 10 days prior to resection

  * Note: patients with DIPG are excluded from the surgical study
* BSA

  * Patients enrolled on dose level -1 must have BSA >= 0.55m2
  * Patients enrolled on dose level -0.5 must have BSA >= 0.75m2
  * Patients enrolled on dose level 0 must have BSA >= 0.55m2
  * Patients enrolled on dose level 1 must have BSA >= 0.75m2
  * Patients enrolled on dose level 2 and 3 must have BSA >= 0.45m2
* Patients must have received prior therapy other than surgery and must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment
* Patients must have received their last dose of known myelosuppressive anticancer therapy at least 21 days prior to enrollment or at least 42 days if nitrosourea
* Biologic or investigational agent (anti-neoplastic): patient must have recovered from any acute toxicity potentially related to the agent and received their last dose of the investigational or biologic agent >= 7 days prior to study enrollment

  * For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur
* Monoclonal antibody treatment and agents with known prolonged half-lives: At least three half-lives must have elapsed prior to enrollment.
* Patients must have had their last fraction of:

  * Craniospinal irradiation (> 24 GRAY [Gy]) or total body irradiation > 12 weeks prior to enrollment
  * Focal irradiation > 2 weeks prior to enrollment
  * >= 3 months since autologous bone marrow/stem cell transplant prior to enrollment
* Neurologic status

  * Patients with neurological deficits should have deficits that are stable for a minimum of 1 week prior to enrollment
  * Patients with seizure disorders may be enrolled if seizures are well controlled on an anti-epileptic drug that is not a strong inducer or inhibitor of CYP3A4/5 are eligible
* Performance status

  * Phase I: Karnofsky performance scale (KPS for > 16 years of age) or Lansky performance score (LPS for =< 16 years of age) assessed within one week of enrollment must be >= 50
  * Surgical study: Karnofsky performance scale (KPS for > 16 years of age) or Lansky performance score (LPS for =< 16 years of age) assessed within one week of enrollment must be >= 60
  * Patients who are unable to walk because of neurologic deficits, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Absolute neutrophil count >= 1.0 x 10^9 cells/ L
* * Platelets >= 100 x 10^9 cells/ L (unsupported, defined as no platelet transfusion within 7 days)
* Hemoglobin >= 8g/dl (unsupported)
* Total bilirubin =< 1.5 times institutional upper limit of normal (ULN)
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) =< 3 x institutional upper limit of normal (ULN)
* Albumin >= 2 g/dl
* Serum creatinine based on age/gender; patients that do not meet the criteria but have a 24 hour creatinine clearance or glomerular filtration rate (GFR) (radioisotope or iothalamate) >= 70 mL/min/1.73 m^2 are eligible
* Patients who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to enrollment
* Patients must be off all colony- forming growth factor(s) for at least 1 week prior to enrollment (i.e. filgrastim, sargramostim or erythropoietin); 2 weeks must have elapsed if patients received long-acting formulations
* Female patients of childbearing potential must have a negative serum or urine pregnancy test
* Patients of childbearing or child fathering potential must be willing to use a medically acceptable form of birth control while being treated on this study; Highly effective contraception methods include:

  * Total abstinence when this is in line with the preferred and usual lifestyle of the patient; periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Combination of any of the two following

    * Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception
    * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository
  * Note: oral contraceptives are allowed but should be used in conjunction with a barrier method of contraception due to unknown effect of drug-drug interaction; in case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment
* Female patients must agree not to breastfeed their infants while on study; patients of child fathering potential (defined as > Tanner stage 2) must use a condom during intercourse while taking the drug during treatment, for 8 weeks after stopping treatment and should not father a child in this period; a condom is required to be used also by vasectomized men during intercourse with a male or female partner in order to prevent delivery of the study drug via semen
* The patient or parent/guardian is able to understand the consent and is willing to sign a written informed consent document according to institutional guidelines; assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Patients who are otherwise deemed clinically unsuitable for surgical resection (applicable for surgical study only)
* Patients who are breast feeding
* Patients with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that would compromise the patient?s ability to tolerate protocol therapy, put them at additional risk for toxicity or would interfere with the study procedures or results
* Patients who are receiving any other anticancer or investigational or/and anti-neoplastic therapies, including chemotherapy, immunotherapy, target therapy, biological response modifiers

  * Previous treatment with CDK4/6 inhibitors (such as PD-0332991, abemaciclib) and/or mTOR inhibitors (such as sirolimus, temsirolimus or everolimus)
  * Patients who are currently receiving treatment with agents that are known to cause corrected QT (QTc) prolongation or induce Torsades de Pointes
  * Known need for major surgery within 14 days of the first dose of ribociclib and everolimus; please note: gastrostomy, insertion of a gastrostomy (G) tube, ventriculo-peritoneal shunt, endoscopic ventriculostomy and central venous access are NOT considered major surgery
* Patient is currently receiving any of the following medications and cannot be discontinued 7 days prior to enrollment:

  * Known strong and moderate inducers or inhibitors of CYP3A4/5, including enzyme inducing anti-convulsant drugs (EIACDs), grapefruit, grapefruit hybrids, pummelos, star-fruit, and Seville oranges
  * Substrates of CYP3A4/5 with a narrow therapeutic index
  * Herbal preparations/medications (except for vitamins) including, but not limited to: St. John?s wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, black cohosh and ginseng; patients should stop using all herbal medications and dietary supplements at least 7 days prior to enrollment
* Clinically significant active cardiac disease, uncontrolled heart disease and/or a history of cardiac dysfunction including any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 12 months prior to screening
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
  * Documented cardiomyopathy
  * Patient has a left ventricular ejection fraction (LVEF) < 50% as determined by echocardiogram (ECHO)
  * History of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality within 12 months of screening
  * Long QT syndrome or known family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:

    * Risk factors for Torsades de Pointe (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia
    * Concomitant use of medication(s) with a known risk to prolong the QT interval and/or days prior to starting study drug) or replaced by safe alternative medication
  * 12-lead electrocardiogram (ECG), any of the following cardiac parameters:

    * QTc > 480 msec
  * Hypertension defined as:

    * Patients 1-17 years of age with blood pressure that is greater than or equal to the 95th percentile for age, height and gender at the time of enrollment; Patients who are ≥ 18 years of age with blood pressure > 140/90 mm of Hg at the time of enrollment.
* Patient is currently receiving warfarin or other coumadin-derived anticoagulant for treatment, prophylaxis or otherwise.
* Patient has a known hypersensitivity to ribociclib or any of its excipients
* Patients with inability to return for required follow-up visits or obtain follow-up studies required to assess toxicity to therapy or to adhere to drug administration plan, other study procedures, and study restrictions.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2018-01-13 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariko D. DeWire-Schottmiller, MD, Principal Investigator — Pediatric Brain Tumor Consortium
Locations (12):
- United States (12):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children Hospital Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - National Cancer Institute Pediatric Oncology Branch, Bethesda, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children Hospital Medical Center, Cincinnati, Ohio
  - Children Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Pediatric Brain Tumor Consortium, Memphis, Tennessee
  - St. Jude Children Research Hospital, Memphis, Tennessee
  - Texas Children's Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is Phase I and Surgical study for children with retinoblastoma protein 1 (Rb1) positive recurrent or refractory central nervous system tumors. Patients were enrolled at Pediatric Brain Tumor Consortium member institutions. The first patient was enrolled on 03/13/2018 and the last patient was enrolled on 11/18/2019. Patients who were enrolled under Surgical study may also be eligible to receive subsequent Phase I defined treatment and evaluable for DLT.
Pre-assignment Details: Total 22 eligible patients were enrolled. 16 of them enrolled on the Phase I study and 6 on the surgical cohort. The 'Started' row includes patients who are eligible for the study. One patient in Phase I dose level 1 withdrew prior to protocol therapy and one patient in Surgical study was not eligible for subsequent protocol therapy. The 'Completed' row includes patients who completed all Phase I protocol therapy or who experienced a protocol defined endpoint which took them off therapy.
Groups:
- Phase I, Dose Level 1: Patients receive ribociclib PO QD on days 1-21 of course 1 and subsequent courses and days 2-21 of course 2 at 120 mg/m2/day, and everolimus PO QD on days 3-28 of course 1 and days 1-28 of subsequent courses at 1.2 mg/m2/day
- Phase I, Dose Level 2: Patients receive ribociclib PO QD on days 1-21 of course 1 and subsequent courses and days 2-21 of course 2 at 170 mg/m2/day, and everolimus PO QD on days 3-28 of course 1 and days 1-28 of subsequent courses at 1.2 mg/m2/day
- Surgical: Patients who are undergoing surgery also received ribociclib PO QD on days 7-10 at 120 mg/m2/day before surgery. Eligible patients were subsequently treated on Phase 1, Dose Level 1.
Period: Overall Study
Arm/Group | Phase I, Dose Level 1 | Phase I, Dose Level 2 | Surgical
Started | 13 | 3 | 5
Received Treatment | 12 | 3 | 5
Completed | 11 | 1 | 5
Not Completed | 2 | 2 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients who are eligible for the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I, Dose Level 1 | Phase I, Dose Level 2 | Surgical | Total
Number analyzed (Participants) | 13 | 3 | 5 | 21
Age, Continuous [Median (Full Range); unit: years] | 10.4 [7.1 to 20.4] | 8.6 [3.9 to 15.9] | 10.8 [7.2 to 17.1] | 10.4 [3.9 to 20.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 1 | 7
  Male | 8 | 2 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 7 | 3 | 3 | 13
  Unknown or Not Reported | 5 | 0 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 8 | 2 | 3 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 13 | 3 | 5 | 21

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Ribociclib and Everolimus
Description: Defined as the highest dose level at which six patients have been treated with at most one patient experiencing a dose limiting toxicity (DLT) and the next higher dose level has been determined to be too toxic. Will be estimated using a Rolling-6 phase I design. Only patients who are evaluable for DLT will be consider for estimating of Maximum Tolerated Dose. Patient who were enrolled under Surgical cohort but received sufficient study defined treatment would also be evaluable for DLT.
Time Frame: 4 weeks
Population: Patients who were evaluable for dose finding assessment were used to determine the MTD. Evaluable patients are those who were eligible, started treatment and either experienced a dose limiting toxicity during course 1 or received adequate amount of treatment and were followed adequately to be assessed for safety during course 1. Evaluable patients could be from either Phase I stratum or from Surgical stratum as long as they received sufficient protocol defined Phase I treatment.
Measure: Number; unit: mg/m^2/day
Groups:
- DLT Evaluable Set: Patients either from Phase I stratum and received treatment from beginning, or from Surgical stratum who subsequently received Phase I defined treatment would be evaluable for MTD as long as they received sufficient Phase I defined treatment. Of the patients enrolled in Phase I stratum, 11 of them were evaluable for dose finding assessment. Of the patients enrolled in Surgical stratum, 5 of them were evaluable for dose finding assessment. Therefore, we have total 16 patients evaluable for dose finding assessment, 11 from Phase I stratum and 5 from Surgical stratum.
Arm/Group | DLT Evaluable Set
Number analyzed (Participants) | 16
mg/m^2/day
  Ribociclib | 120
  Everolumus | 1.2

2. Primary Outcome: Average Tumor and Plasma Concentrations of Ribociclib for the Surgical Study
Description: Average tumor Ribociclib concentrations will be compared to plasma concentrations. The mean tumor-to-plasma ratio of Ribociclib at the time of surgery will be described.
Time Frame: Surgical study: Prior to starting ribociclib (day -7 or -10), prior to ribociclib dose on days -5 & -2, day 0, and at the time of surgery
Population: Patients who were enrolled on surgical study and with tumor and matching plasma samples available.
Measure: Median (Full Range); unit: ratio
Groups:
- Surgical: Patients who are undergoing surgery also receive ribociclib PO QD on days 7-10 at 120 mg/m2/day before surgery
Arm/Group | Surgical
Number analyzed (Participants) | 5
ratio | 14.6 [2.22 to 53.4]

3. Secondary Outcome: Objective Responses (Complete Response + Partial Response)
Description: Number of patients with sustained objective responses will be reported by stratum and dose. Objective response refers to at least 50% reduction in 2 dimensional measurements of the tumor. In order to count towards this objective, any response needs to be sustained for at least 8 weeks.
Time Frame: Up to 2 years
Population: Patients who received Phase I treatment were included in the analysis. One patient in Phase I study withdrew prior to beginning protocol therapy and one patient in Surgical study was not eligible to start Phase I treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I, Dose Level 1 | Phase I, Dose Level 2 | Surgical
Number analyzed (Participants) | 12 | 3 | 5
Participants | 0 | 0 | 0

4. Secondary Outcome: Percent Change in ki67 Between Archival and Post-treatment Tissue
Description: For the surgical study, Ki67 will be evaluated in paired pre-treatment tumor (diagnostic) and post-treatment tumor (recurrent) tissue in consenting patients to assess percent change. The percent of Ki67 in tumor tissues will be measured and the result is presented as the percent of Ki67 in post-treatment tumor minus the percent of Ki67 measured in pre-treatment tumor.
Time Frame: Up to 2 years
Population: Consented patients in surgical study with pre-treatment tumor and post-treatment tumor tissue available
Measure: Median (Full Range); unit: Change of Percentage of Ki67 in Tumor
Arm/Group | Surgical
Number analyzed (Participants) | 2
Change of Percentage of Ki67 in Tumor | -20 [-35 to -5]

5. Other Pre Specified Outcome: Ribociclib AUC (Area Under the Plasma Concentration Versus Time Curve) as Obtained From the Patients Who Received Phase I Defined Treatment
Description: Ribociclib plasma concentration-time data obtained from patients who received Phase I defined treatment will be modeled using compartmental approaches to estimate the AUC (hr*μM) for each dose level on days 1 and 17 of course 1. Patients who were enrolled in the Surgical stratum but subsequently received Phase I defined treatment with PK data available will also be included in the analysis population. 5 patients from surgical stratum received dose level 1 treatment.
Time Frame: Pre-dose, 1, 2, 4, 8, 24, 32 (day 1 course 1 only), & 48 (day 1 course 1 only) hours after dose on days 1 and 17 of course 1.
Population: Patients with blood samples collected for pharmacokinetic studies on days 1 and 17 of course 1 were included. Surgical patients who received Phase I treatment with samples collected were also included in Dose Level 1. There are total 17 patients received dose level 1 treatment and 3 patients received dose level 2 treatment.
Measure: Median (Full Range); unit: hr*uM
Groups:
- Dose Level 1, Day 1 of Course 1: Patients receive ribociclib PO QD on days 1-21 of course 1 and subsequent courses and days 2-21 of course 2 at 120 mg/m2/day, and everolimus PO QD on days 3-28 of course 1 and days 1-28 of subsequent courses at 1.2 mg/m2/day. Samples are collected on Day 1 of Course 1.
- Dose Level 1, Day 17 of Course 1: Patients receive ribociclib PO QD on days 1-21 of course 1 and subsequent courses and days 2-21 of course 2 at 120 mg/m2/day, and everolimus PO QD on days 3-28 of course 1 and days 1-28 of subsequent courses at 1.2 mg/m2/day. Samples are collected on Day 17 of Course 1.
- Dose Level 2, Day 1 of Course 1: Patients receive ribociclib PO QD on days 1-21 of course 1 and subsequent courses and days 2-21 of course 2 at 170 mg/m2/day, and everolimus PO QD on days 3-28 of course 1 and days 1-28 of subsequent courses at 1.2 mg/m2/day. Samples are collected on Day 1 of Course 1.
- Dose Level 2, Day 17 of Course 1: Patients receive ribociclib PO QD on days 1-21 of course 1 and subsequent courses and days 2-21 of course 2 at 170 mg/m2/day, and everolimus PO QD on days 3-28 of course 1 and days 1-28 of subsequent courses at 1.2 mg/m2/day. Samples are collected on Day 17 of Course 1
Arm/Group | Dose Level 1, Day 1 of Course 1 | Dose Level 1, Day 17 of Course 1 | Dose Level 2, Day 1 of Course 1 | Dose Level 2, Day 17 of Course 1
Number analyzed (Participants) | 16 | 15 | 3 | 2
hr*uM | 3.96 [2.6 to 11.2] | 10.3 [5.3 to 18.7] | 12.0 [5.4 to 13.4] | 10.15 [9.6 to 10.7]

6. Other Pre Specified Outcome: Everolimus AUC (Area Under the Plasma Concentration Versus Time Curve) as Obtained From the Phase I Study
Description: Everolimus plasma concentration-time data obtained from patients who received Phase I defined treatment will be modeled using compartmental approaches to estimate the AUC (hr*nM) for each dose level on day 17 of course 1 and day 1 of course 2. Patients who were enrolled in the Surgical stratum but subsequently received Phase I defined treatment with PK data available will also be included in the analysis population. 5 patients from surgical stratum received dose level 1 treatment.
Time Frame: Pre-dose, 0.5 (course 2 only), 1, 1.5 (course 2 only), 2, 4, 6 (course 2 only), 8, 24 hours after dose on day 17 of course 1, and day 1 of course 2.
Population: Patients with blood samples collected for pharmacokinetic studies on day 17 of course 1 and day 1 of course 2 were included. Surgical patients who received Phase I treatment with samples collected were also included in Dose Level 1. There are total 17 patients received dose level 1 treatment and 3 patients received dose level 2 treatment. Analysis population only includes treated patients with corresponding PK data available.
Measure: Median (Full Range); unit: hr*nM
Groups:
- Dose Level 1, Day 1 of Course 2: Patients receive ribociclib PO QD on days 1-21 of course 1 and subsequent courses and days 2-21 of course 2 at 120 mg/m2/day, and everolimus PO QD on days 3-28 of course 1 and days 1-28 of subsequent courses at 1.2 mg/m2/day. Samples are collected on Day 1 of Course 2.
- Dose Level 2, Day 1 of Course 2: Patients receive ribociclib PO QD on days 1-21 of course 1 and subsequent courses and days 2-21 of course 2 at 170 mg/m2/day, and everolimus PO QD on days 3-28 of course 1 and days 1-28 of subsequent courses at 1.2 mg/m2/day. Samples are collected on Day 1 of Course 2.
Arm/Group | Dose Level 1, Day 17 of Course 1 | Dose Level 1, Day 1 of Course 2 | Dose Level 2, Day 17 of Course 1 | Dose Level 2, Day 1 of Course 2
Number analyzed (Participants) | 14 | 10 | 2 | 2
hr*nM | 201 [52.7 to 399] | 80.1 [29.8 to 146] | 147.5 [119 to 176] | 59 [42.5 to 75.5]

7. Other Pre Specified Outcome: Ribociclib Half-Life as Obtained From the Phase 1 Study
Description: Ribociclib plasma concentration-time data obtained from patients received Phase I defined treatment will be modeled using compartmental approaches to estimate the half-life (hrs) for each dose level on days 1 and 17 of course 1. Patients who were enrolled in the Surgical stratum but subsequently received Phase I defined treatment with PK data available will also be included in the analysis population. 5 patients from surgical stratum received dose level 1 treatment.
Time Frame: as for outcome 5
Population: Patients with blood samples collected for pharmacokinetic studies on days 1 and 17 of course 1 were included. Surgical patients who received Phase I treatment with samples collected were also included in Dose Level 1. There are total 17 patients received dose level 1 treatment and 3 patients received dose level 2 treatment. The analysis population only includes patients with corresponding PK data available at that timepoint.
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Level 1, Day 1 of Course 1 | Dose Level 1, Day 17 of Course 1 | Dose Level 2, Day 1 of Course 1 | Dose Level 2, Day 17 of Course 1
Number analyzed (Participants) | 16 | 15 | 3 | 2
hours | 11.7 [8.0 to 18.0] | 8.9 [7.3 to 17.3] | 8.5 [8.4 to 13.9] | 7.5 [5.5 to 9.5]

8. Other Pre Specified Outcome: Everolimus Half Life as Obtained From the Phase 1 Study
Description: Everolimus plasma concentration-time data obtained from patients received Phase I defined treatment will be modeled using compartmental approaches to estimate the half-life (hrs) for each dose level on day 17 of course 1 and day 1 of course 2. Patients who were enrolled in the Surgical stratum but subsequently received Phase I defined treatment with PK data available will also be included in the analysis population. 5 patients from surgical stratum received dose level 1 treatment.
Time Frame: Pre-dose, 0.5 (course 2 only), 1, 1.5 (course 2 only), 2, 4, 6 (course 2 only), 8, & 24 hours after dose on day 17 of course 1, and day 1 of course 2
Population: Patients with blood samples collected for pharmacokinetic studies on day 17 of course 1 and day 1 of course 2 were included. Surgical patients who received Phase I treatment with samples collected were also included in Dose Level 1. There are total 17 patients received dose level 1 treatment and 3 patients received dose level 2 treatment. The analysis population only includes patients with corresponding PK data available at that timepoint.
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Level 1, Day 17 of Course 1 | Dose Level 1, Day 1 of Course 2 | Dose Level 2, Day 17 of Course 1 | Dose Level 2, Day 1 of Course 2
Number analyzed (Participants) | 14 | 10 | 2 | 2
hours | 13.5 [8.5 to 23.1] | 14.5 [6.9 to 23.9] | 11.2 [9.0 to 13.3] | 11.5 [7.3 to 15.6]

ADVERSE EVENTS:
Time Frame: Up to 2 years after starting treatment
Description: Adverse events (AEs) were graded using CTCAE v5.0. AEs collected per protocol included: a) grade 1 and 2 AEs if attribution was at least possibly related to Ribociclib or Everolimus and b) all grade 3+ AEs on treatment and within 30 days off treatment. AEs were summarized in SAE and Other AE tables below. All mortality on this study were due to disease. Two patients did not started phase I protocol defined therapy and were not counted as at risk.
Arm/Group | Phase I, Dose Level 1 | Phase I, Dose Level 2 | Surgical
All-Cause Mortality (participants affected / at risk) | 5/12 | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 6/12 | 1/3 | 1/5
Other Adverse Events (participants affected / at risk) | 12/12 | 3/3 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Dose Level 1 (N=12) | Phase I, Dose Level 2 (N=3) | Surgical (N=5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Disease progression (General disorders) | 2 (2) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
DECREASED VISUAL FIELDS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Edema cerebral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Glossopharyngeal nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
MOTOR APRAXIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 2 (4) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Dose Level 1 (N=12) | Phase I, Dose Level 2 (N=3) | Surgical (N=5)
Anemia (Blood and lymphatic system disorders) | 4 (6) | 1 (11) | 4 (8)
Corneal ulcer (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 4 (7) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (6) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (6) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 6 (8) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (5) | 2 (13) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (8) | 0 (0)
Cholesterol high (Investigations) | 4 (5) | 2 (3) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (9) | 3 (9) | 4 (13)
Neutrophil count decreased (Investigations) | 5 (11) | 2 (6) | 5 (11)
Platelet count decreased (Investigations) | 3 (3) | 1 (1) | 2 (10)
Weight gain (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 2 (7) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 6 (15) | 3 (8) | 4 (18)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (4)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3) | 1 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
DISEASE PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (5) | 0 (0) | 0 (0)
PEDIATRIC HYPERTENSION (Vascular disorders) | 0 (0) | 2 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator Initiated Interventional Trial Agreement between Novartis and PBTC and Cincinnati Children's Hospital Medical Center.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/20/NCT03387020/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/20/NCT03387020/ICF_001.pdf